CLINICAL TRIAL: NCT01844180
Title: A Phase 2, Multi-center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ONO-2952 in Female Subjects With Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D)
Brief Title: A Phase 2, Multi-center Study to Evaluate the Efficacy and Safety of ONO-2952 in Female Subjects With Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D)
Acronym: RESTORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-2952POU004
Record Dates: First submitted 2013-04-24; First posted 2013-05-01 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Irritable Bowel Syndrome; IBS; ONO-2952
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — ONO-2952

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental Arm 1 (Experimental): ONO-2952 low dose every day for 4 weeks
  Interventions: Drug: ONO-2952
- Experimental Arm 2 (Experimental): ONO-2952 high dose every day for 4 weeks
  Interventions: Drug: ONO-2952
- Placebo Arm (Placebo Comparator): ONO-2952 Matching Placebo every day for 4 weeks
  Interventions: Drug: ONO-2952 Matching Placebo

INTERVENTIONS:
Drug: ONO-2952
  Arms: Experimental Arm 1; Experimental Arm 2
Drug: ONO-2952 Matching Placebo
  Arms: Placebo Arm

SUMMARY:
The objective of this study is to explore efficacy, safety and tolerability of ONO-2952 in female subjects with Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D).

ELIGIBILITY:
Inclusion Criteria:

1. Female 18-65 years of age (inclusive)
2. Diagnosed with IBS based on the following criteria (Rome III criteria):

   * Symptom onset at least 6 months prior to diagnosis, and
   * Recurrent abdominal pain or discomfort at least 3 days per month for the past 3 months, and
   * Abdominal discomfort or pain associated with two or more of the following at least 25% of the time:

     1. Improvement with defecation
     2. Onset associated with a change in frequency of stool/defecation
     3. Onset associated with a change in form (appearance) of stool
3. Diagnosed with IBS-D, defined as loose/watery stools ≥ 25% and hard/lumpy stools ≤ 25% of defecations

Exclusion Criteria:

* Any structural abnormality of the gastrointestinal (GI) tract (other than esophagitis or gastritis)
* History of Crohn's disease, ulcerative colitis, diabetes mellitus, lactose malabsorption, malabsorption syndromes, celiac sprue, or any upper GI symptoms that may impact the assessment of IBS symptoms

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Abdominal pain or stool symptoms in female subjects with IBS-D by using a numeric pain rating scale and the Bristol Stool Scale (BSS) | 4 weeks

SECONDARY OUTCOMES:
Change in IBS related symptoms and quality of life (QoL) by questionaire assessments | 4 weeks
Safety assessed through adverse events and clinical laboratory values | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (48):
- United States (48):
  - Anniston Clinical Site, Anniston, Alabama
  - Goodyear Clinical Site, Goodyear, Arizona
  - Tucson Clinical Site, Tucson, Arizona
  - North Little Rock Clinical Site, North Little Rock, Arkansas
  - Carlsbad Clinical Site, Carlsbad, California
  - San Diego Clinical Site, San Diego, California
  - Boynton Beach Clinical Site, Boynton Beach, Florida
  - Clearwater Clinical Site, Clearwater, Florida
  - Deland Clinical Site, DeLand, Florida
  - Hialeah Clinical Site, Hialeah, Florida
  - Lauderdale Lakes Clinical Site, Lauderdale Lakes, Florida
  - Orlando Clinical Site, Orlando, Florida
  - Port Orange Clinical Site, Port Orange, Florida
  - South Miami Clinical Site, South Miami, Florida
  - St. Petersburg Clinical Site, St. Petersburg, Florida
  - Tampa Clinical Site, Tampa, Florida
  - West Palm Clinical Site, West Palm, Florida
  - Oak Lawn Clinical Site, Oak Lawn, Illinois
  - Wichita Clinical Site, Wichita, Kansas
  - New Orleans Clinical Site, New Orleans, Louisiana
  - Chesterfield Clincial Site, Chesterfield, Michigan
  - Billings Clinical Site, Billings, Montana
  - Reno Clinical Site, Reno, Nevada
  - Lebanon Clinical Site, Lebanon, New Hampshire
  - Albuquerque Clinical Site, Albuquerque, New Mexico
  - Great Neck Clinical Site, Great Neck, New York
  - Cary Clinical Site, Cary, North Carolina
  - Highpoint Clinical Site, Highpoint, North Carolina
  - Raleigh Clinical Site, Raleigh, North Carolina
  - Winston-Salem Clinical Site, Winston-Salem, North Carolina
  - Akron Clinical Site, Akron, Ohio
  - Columbus Clinical Site, Columbus, Ohio
  - Dayton Clinical Site, Dayton, Ohio
  - Groveport Clinical Site, Groveport, Ohio
  - Mentor Clinical Site, Mentor, Ohio
  - Norman Clinical Site, Norman, Oklahoma
  - Lansdale Clinical Site, Landsdale, Pennsylvania
  - Greer Clinical Site, Greer, South Carolina
  - Mt. Pleasant Clinical Site, Mt. Pleasant, South Carolina
  - Chattanooga Clinical Site, Chattanooga, Tennessee
  - Germantown Clinical Site, Germantown, Tennessee
  - Pasadena Clinical Site, Pasadena, Texas
  - Plano Clinial Site, Plano, Texas
  - San Antonio Clinical Site, San Antonio, Texas
  - Logan Clinical Site, Logan, Utah
  - Ogden Clinical Site, Ogden, Utah
  - Salt Lake City Clinical Site, Salt Lake City, Utah
  - Sandy Clinical Site, Sandy City, Utah

REFERENCES:
- [Derived] Whitehead WE, Duffy K, Sharpe J, Nabata T, Bruce M. Randomised clinical trial: exploratory phase 2 study of ONO-2952 in diarrhoea-predominant irritable bowel syndrome. Aliment Pharmacol Ther. 2017 Jan;45(1):14-26. doi: 10.1111/apt.13839. Epub 2016 Nov 7. PMID 27910150